CLINICAL TRIAL: NCT06457672
Title: Assessment of The Accuracy of Complete Crown 3D Superimposition Technique Relative to The Gold Standard Technique for Digital Quantification of Volumetric Soft Tissue Changes in The Esthetic Zone
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: British University In Egypt (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Hassan, assistant lecturer, British University In Egypt
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CU1612
Record Dates: First submitted 2024-06-09; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- group I (Experimental): complete crown technique for superimposition of digital models
  Interventions: Diagnostic Test: Group I; Diagnostic Test: Group II

INTERVENTIONS:
Diagnostic Test: Group I — Complete Crown technique of superimposition
Diagnostic Test: Group II — Gold standard technique of superimposition

SUMMARY:
The aim of this study is to assess the precision of the complete crown technique employed for the superimposition of 3D models, specifically in the quantitative volumetric evaluation of gingival tissues. This technique was initially introduced in an in-vitro study by Dritsas et al. (2023) as a means to achieve an accurate, reproducible, and simple method for quantification of gingival recession.

DETAILED DESCRIPTION:
This study will involve the analysis of digital models in. ply format acquired through intraoral scanning of patients scheduled for esthetic crown lengthening,

A. Pre-analytical Phase:

In an interview, a full medical history is obtained. Clinical and radiographic examinations are completed before consent signing for study enrollment.

Full mouth supra and subgingival debridement will be performed for patients using an ultrasonic device with supragingival scaling inserts, followed by Universal or Gracey's curettes for thorough subgingival debridement. Patient preparation will be completed in a single visit. Comprehensive oral hygiene instructions will be provided to the patient, including instructions for brushing teeth twice daily using a soft toothbrush and employing a circular scrub technique.

Additionally, guidance will be given on interdental cleansing, using either waxed dental floss or a toothpick appropriate for the size of the interdental embrasure.

Surgical procedure:

After a period of 4-6 weeks from the initial therapy, patients will be recalled. After ensuring the fulfillment of all inclusion criteria, they will be scheduled for surgery.

Following local anesthesia, the surgical procedure will be initiated with demarcation of CEJ position on the mid-buccal aspect of the teeth. The width of the central incisors will be identified by measuring the teeth width at the level of interproximal contact using UNC periodontal probe. Then the ideal tooth length will be calculated through the central tooth width to length ratio of 75-85%. The canines will be marked at the same level as the central incisors while the lateral incisors will be marked at 1 mm apical to the central incisors. Zenith points will be marked using a tissue pen at 1 mm distally shifted to the midline of centrals, 0.4 mm distally on the laterals, and mostly on the midline of canines (Chu et al., 2009). The interdental papillae levels will be evaluated. If they are situated at a level higher than the half of the adjacent tooth crown, then they will need to be shortened and will be included in the cutting design. If the interdental papillae levels are equal to or less than half the length of the adjacent tooth crown, then the cutting lines will be thinned from the zenith points to the papillae tips (Spear et al., 2006).

An internal bevel incision using #15c blade will be performed following the anatomy of the CEJ. The incision will be made at 45 degrees to the bone at each tooth, preserving the interdental papillae when needed. This will be followed by an intra-sulcular incision in order to remove the strip of the outlined marginal gingiva.

When bone removal is advocated, a full-thickness flap will be elevated to the level of the alveolar bone crest exposing 2-3 mm of bone using a normal mucoperiosteal elevator(Arora et al., 2013). The cementoenamel junction-alveolar bone crest (CEJ-ABC) distance will be measured on the mid-buccal aspect. Then, ostectomy and osteoplasty will be performed using an end-cutting bur and round bur, aiming to attain a 2 mm CEJ-ABC distance for attaining a normal biological width.

Finally, the flap will be repositioned, and simple interrupted sutures of 4/0 vicryl will be used to keep the papillae in place, using a normal needle holder(Palomo & Kopczyk, 1978;Deas et al., 2004).

B. Analytical phase:

Each model will go through a trimming process utilizing the arch cut tool. Subsequently, a base will be created for each model employing the model base tool. A thorough inspection is performed to identify any potential voids in the model base. In cases where voids are detected, the "fill holes" tool will be employed to rectify and fill any voids present within the model base. Implementation of the superimposition: Utilizing the superimposition tool, an initial manual alignment of the digital models will be performed, followed by the superimposition procedure. The T0 model will be designated as the reference model, while the first T6 model will be chosen as the moving model. The second T6 model will be designated as the moving.001 model.

For the complete crown technique, the crown of the tooth corresponding to the gingival margin under evaluation will be selected using the paint method and circular selection tool. The same selection process will be applied to the moving model. In the case of the gold standard technique, adjacent intact teeth and a portion of the palatal gingiva will be selected. Superimpositions will be executed utilizing the software's iterative closest point algorithm (ICP). A heat map will be generated to verify the accuracy of the superimposition process.

Superimposition accuracy:

Models will be exported in superimposed orientations to the Geomagic software6 for the measurement of superimposition accuracy, specifically the root mean square of the tooth corresponding to the gingival margin where volumetric changes are of interest, using the 3D compare tool in Geomagic software.

Marginal and Volumetric changes:

For assessing changes at the gingival margin level, all three models will be selected, and a cross section will be generated at the center of the targeted tooth, followed by linear measurements.

To evaluate volumetric changes, a Boolean modifier will be applied between the T0 model and the T6 model. Excess mesh vertices will then be removed using the clean model tool. Subsequently, the excised gingival margin will become readily apparent and quantifiable, allowing for the measurement of its volume through the utilization of the 3D print module within the BlenderForDental software.

C.Post-analytical Phase:

The evaluation will be conducted by two periodontists possessing varying levels of experience.

Subsequently, inter-observer agreements will be quantified. To assess intra-observer agreement, one of the two periodontists will perform the evaluation on two occasions, with a two-week interval between each assessment (Vasilakos et al., 2017).

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years or older.
2. Patients requiring esthetic crown lengthening.
3. Full-mouth plaque and bleeding score not exceeding 20%.
4. Presence of at least 2.5 mm keratinized tissue width (Pontoriero & Carnevale, 2001).
5. Patients showing motivation to comply with post-operative care instructions and follow-up appointments.

Exclusion Criteria:

1. Systemic health conditions that contraindicate or affect healing of periodontal surgery.
2. Patients requiring prosthetic crowns or restorations in the esthetic zone.
3. Gummy smile with normal tooth proportions.
4. Patients treated with medications known to affect the gingiva (Phenytoin, Cyclosporine and Nifedipine).
5. Smokers.
6. Pregnant and nursing females.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Superimposition accuracy | 6 months
  Using Geomagic Software (RMS) in Millimeter(mm)

SECONDARY OUTCOMES:
Soft tissue volumetric Changes | 6 months
  Digital using intraoral scanner and blenderfordental software in Millimeter(mm)
Gingival Margin level change | 6 months
  Digital using intraoral scanner and blenderfordental software in Millimeter(mm)
Intra-Inter Assessor reliability | 6 months
  Intraclass correlation coefficient
Operator's satisfaction | 6 months
  Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Hassan, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided